CLINICAL TRIAL: NCT00869908
Title: The Effect of NovoMix® 30, Levemir® or NovoRapid® (Alone or in Combination) in Subjects With Type 2 Diabetes Previously Treated With Other Anti-diabetic Medication. A 24-week, International, Prospective, Multi-centre, Open-labelled, Non-interventional Study
Brief Title: Observational Study on the Effect of NovoMix® 30, Levemir® or NovoRapid® (Alone or Combined) in Type 2 Diabetics Previously Treated With Anti-diabetic Medication
Acronym: A1chieve®
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3693
Record Dates: First submitted 2009-03-23; First posted 2009-03-26 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Detemir; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin aspart; Drug: insulin detemir; Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: NovoRapid®; ANA
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
Drug: biphasic insulin aspart — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation

SUMMARY:
This study is conducted in Africa, Asia, South America and Europe. The aim of this observational study is to document the experience with the study insulins when used in routine clinical practice. After the physician's decision to start insulin treatment using NovoMix® 30, Levemir® or NovoRapid® (alone or combined), type 2 diabetics will be eligible to be included in this study at the physician's discretion

ELIGIBILITY:
Inclusion Criteria:

* After the physician has taken the decision to use NovoMix®30, Levemir® or NovoRapid® (alone or combined), any subject with type 2 diabetes who is not treated with these insulins or who has started on these insulin within the last 4 weeks before inclusion into this study is eligible for the study.
* The selection of the subjects will be at the discretion of the individual physician.

Exclusion Criteria:

* Subjects treated with NovoMix® 30, Levemir® or NovoRapid® (alone or in combination) for more than 4 weeks before inclusion into this study.
* Subjects who were previously enrolled in this study.
* Subjects with a hypersensitivity to NovoMix® 30, Levemir® or NovoRapid® or to any of the excipients.
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within the next 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only people with type 2 diabetes treated by general practitioners and specialists who prescribe insulin analogues in their routine practice will be included
Sampling Method: Non-Probability Sample
Enrollment: 66726 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse drug reactions and major hypoglycaemic events reported as serious adverse drug reactions | at baseline, 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Evaluate the prescribing patterns and choice of insulin analogues in routine clinical practice | at baseline, 12 weeks and 24 weeks
Change in number of hypoglycaemic events | at baseline, 12 weeks and 24 weeks
Change in HbA1c | at baseline, 12 weeks and 24 weeks
Change in FPG (Fasting Plasma Glucose) | at baseline, 12 weeks and 24 weeks
Change in PPG (postprandial glucose) | at baseline, 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (22):
- Novo Nordisk Investigational Site, Algiers, Algeria
- Novo Nordisk Investigational Site, Prov. de Buenos Aires, Argentina
- Novo Nordisk Investigational Site, Dhaka, Bangladesh
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China
- Novo Nordisk Investigational Site, Cairo, Egypt
- Novo Nordisk Investigational Site, Bangalore, India
- Novo Nordisk Investigational Site, Jakarta, Indonesia
- Novo Nordisk Investigational Site, Tehran, Iran
- Novo Nordisk Investigational Site, Amman, Jordan
- Novo Nordisk Investigational Site, Tripoli, Libya
- Novo Nordisk Investigational Site, Selangor Darul Ehsan, Malaysia
- Novo Nordisk Investigational Site, Mexico City, Mexico
- Novo Nordisk Investigational Site, Casablanca, Morocco
- Novo Nordisk Investigational Site, Karachi, Pakistan
- Novo Nordisk Investigational Site, Manila, Philippines
- Novo Nordisk Investigational Site, Moscow, Russia
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Singapore, Singapore
- Novo Nordisk Investigational Site, Seoul, South Korea
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Novo Nordisk Investigational Site, Tunisia, Tunisia
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Home P, Naggar NE, Khamseh M, Gonzalez-Galvez G, Shen C, Chakkarwar P, Wenying Y. An observational non-interventional study of people with diabetes beginning or changed to insulin analogue therapy in non-Western countries: the A1chieve study. Diabetes Res Clin Pract. 2011 Dec;94(3):352-63. doi: 10.1016/j.diabres.2011.10.021. PMID 22153567
- [Result] Shah S, Zilov A, Malek R, Soewondo P, Bech O, Litwak L. Improvements in quality of life associated with insulin analogue therapies in people with type 2 diabetes: results from the A1chieve observational study. Diabetes Res Clin Pract. 2011 Dec;94(3):364-70. doi: 10.1016/j.diabres.2011.10.020. PMID 22153568
- [Result] Shah SN, Litwak L, Haddad J, Chakkarwar PN, Hajjaji I. The A1chieve study: a 60 000-person, global, prospective, observational study of basal, meal-time, and biphasic insulin analogs in daily clinical practice. Diabetes Res Clin Pract. 2010 May;88 Suppl 1:S11-6. doi: 10.1016/S0168-8227(10)70003-6. PMID 20466163
- [Result] Randeree H, Liebl A, Hajjaji I, Khamseh M, Zajdenverg L, Chen JW, Haddad J. Safety and effectiveness of bolus insulin aspart in people with type 2 diabetes: a1chieve sub-analysis. Diabetes Ther. 2013 Jun;4(1):153-66. doi: 10.1007/s13300-013-0026-y. Epub 2013 Jun 12. PMID 23757032
- [Result] Zilov A, El Naggar N, Shah S, Shen C, Haddad J. Insulin detemir in the management of type 2 diabetes in non-Western countries: safety and effectiveness data from the A(1)chieve observational study. Diabetes Res Clin Pract. 2013 Sep;101(3):317-25. doi: 10.1016/j.diabres.2013.06.003. PMID 24119589
- [Result] Shah S, Yang W, Hasan MI, Malek R, Molskov Bech O, Home P. Biphasic insulin aspart 30 in insulin-naive people with type 2 diabetes in non-western nations: results from a regional comparative multinational observational study (A(1)chieve). Diabetes Technol Ther. 2013 Nov;15(11):954-63. doi: 10.1089/dia.2013.0074. Epub 2013 Sep 20. PMID 24053450
- [Result] Home PD, Latif ZA, Gonzalez-Galvez G, Prusty V, Hussein Z. The effectiveness and safety of beginning insulin aspart together with basal insulin in people with type 2 diabetes in non-Western nations: results from the A(1)chieve observational study. Diabetes Res Clin Pract. 2013 Sep;101(3):326-32. doi: 10.1016/j.diabres.2013.06.005. PMID 24119590
- [Result] Litwak L, Goh SY, Hussein Z, Malek R, Prusty V, Khamseh ME. Prevalence of diabetes complications in people with type 2 diabetes mellitus and its association with baseline characteristics in the multinational A1chieve study. Diabetol Metab Syndr. 2013 Oct 24;5(1):57. doi: 10.1186/1758-5996-5-57. PMID 24228724
- [Result] Chen L, Xing X, Lei M, Liu J, Shi Y, Li P, Qin G, Li C, Li Y, Wang Q, Gao T, Hu L, Wang Y, Yang W. Biphasic insulin aspart 30 improved glycemic control in Chinese patients with type 2 diabetes poorly controlled on oral glucose-lowering drugs: a subgroup analysis of the A(1)chieve study. Chin Med J (Engl). 2014;127(2):208-12. PMID 24438605
- [Result] Hwang YC, Kang JG, Ahn KJ, Cha BS, Ihm SH, Lee S, Kim M, Lee BW. The glycemic efficacies of insulin analogue regimens according to baseline glycemic status in Korean patients with type 2 diabetes: sub-analysis from the A(1)chieve((R)) study. Int J Clin Pract. 2014 Nov;68(11):1338-44. doi: 10.1111/ijcp.12482. Epub 2014 Oct 6. PMID 25284679
- [Result] Yang W, Zhuang X, Li Y, Wang Q, Bian R, Shen J, Hammerby E, Yang L. Improvements in quality of life associated with biphasic insulin aspart 30 in type 2 diabetes patients in China: results from the A1chieve(R) observational study. Health Qual Life Outcomes. 2014 Nov 26;12:137. doi: 10.1186/s12955-014-0137-9. PMID 25424627
- [Result] Khamseh ME, Haddad J, Yang W, Zilov A, Bech OM, Hasan MI. Safety and effectiveness of biphasic insulin aspart 30 in different age-groups: a1chieve sub-analysis. Diabetes Ther. 2013 Dec;4(2):347-61. doi: 10.1007/s13300-013-0033-z. Epub 2013 Jul 17. PMID 23860823
- [Result] Home PD, Shen C, Hasan MI, Latif ZA, Chen JW, Gonzalez Galvez G. Predictive and explanatory factors of change in HbA1c in a 24-week observational study of 66,726 people with type 2 diabetes starting insulin analogs. Diabetes Care. 2014;37(5):1237-45. doi: 10.2337/dc13-2413. Epub 2014 Mar 4. PMID 24595628
- [Result] El-Naggar N, Almansari A, Khudada K, Salman S, Mariswamy N, Abdelfattah W, Hashim F. The A1 chieve study - an observational non-interventional study of patients with type 2 diabetes mellitus initiating or switched to insulin analogue therapy: subgroup analysis of the Gulf population. Int J Clin Pract. 2013 Feb;67(2):128-38. doi: 10.1111/ijcp.12078. PMID 23305475
- [Result] El Naggar NK, Soewondo P, Khamseh ME, Chen JW, Haddad J. Switching from biphasic human insulin 30 to biphasic insulin aspart 30 in type 2 diabetes is associated with improved glycaemic control and a positive safety profile: results from the A(1)chieve study. Diabetes Res Clin Pract. 2012 Dec;98(3):408-13. doi: 10.1016/j.diabres.2012.09.043. PMID 23217267
- [Derived] Song SO, Hwang YC, Ahn KJ, Cha BS, Song YD, Lee DW, Lee BW. Clinical Characteristics of Patients Responding to Once-Daily Basal Insulin Therapy in Korean Subjects with Type 2 Diabetes. Diabetes Ther. 2015 Dec;6(4):547-558. doi: 10.1007/s13300-015-0140-0. Epub 2015 Oct 29. PMID 26515457
- [Derived] Gupta V, Baabbad R, Hammerby E, Nikolajsen A, Shafie AA. An analysis of the cost-effectiveness of switching from biphasic human insulin 30, insulin glargine, or neutral protamine Hagedorn to biphasic insulin aspart 30 in people with type 2 diabetes. J Med Econ. 2015 Apr;18(4):263-72. doi: 10.3111/13696998.2014.991791. Epub 2015 Jan 2. PMID 25426701
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com